CLINICAL TRIAL: NCT03495986
Title: Spinal Cord Injury Exercise and Nutrition Conceptual Engagement (SCIENCE)
Brief Title: Spinal Cord Injury Exercise and Nutrition Conceptual Engagement
Acronym: SCIENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Eduard Tiozzo, PhD, Research Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190659; R01HD091278-01 (NIH); 6996 (Other: Pennsylvania State University)
Record Dates: First submitted 2018-03-02; First posted 2018-04-12 (Actual); Results first posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injuries; Metabolic Syndrome; Dietary Modification; Paraplegia; Tetraplegia
Keywords: Functional Electrical Stimulation; Exercise; Body Composition
MeSH Terms: conditions — Spinal Cord Injuries; Metabolic Syndrome; Paraplegia; Quadriplegia; Motor Activity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Home-Based Exercise & Diet Group (Experimental): 16-week home based functional electrical stimulation leg cycle ergometry exercise program and diet intervention
  Interventions: Device: Functional Electrical Stimulation Leg Cycle Ergometry; Behavioral: Diet
- Home-Based Diet Alone Group (Placebo Comparator): Diet intervention
  Interventions: Behavioral: Diet

INTERVENTIONS:
Device: Functional Electrical Stimulation Leg Cycle Ergometry — Exercise training will consist of three to five, 40-67 minute sessions (200 minutes at target intensity) each week for a total of 16 weeks at 70% maximal heart rate; 10-minute warm-up and cool-down sessions will accompany each exercise session.
  Arms: Home-Based Exercise & Diet Group
Behavioral: Diet — An individualized, detailed dietary plan consistent with My Healthy Plate Dietary Guidelines of America will be followed under supervision of Registered Dietitian with weekly telemedicine conferences and monitored dietary intake via MyFitnessPal.

SUMMARY:
Evaluate and compare the health benefits of an at home exercise program using functional electrical stimulation (FES) for lower extremity exercise with diet versus a diet alone group in adults with spinal cord injury.

DETAILED DESCRIPTION:
The purpose of this proposal is to evaluate and compare the health benefits of home-based functional electrical stimulation leg cycle ergometry plus diet (HBFESLCE + Diet) to home-based (HB) Diet alone. This is a randomized, baseline-controlled, prospective, interventional trial to assess the impact of a 16-week exercise and/or diet intervention on selected fitness parameters in adults with high SCI. Primary outcome measures will include body composition by iDXA, insulin sensitivity, glucose effectiveness and BMR, while secondary outcomes will include lower extremity BMC and density, lipid profiles, and hsCRP determined before and after the 16-week interventions. Subjects will be randomly assigned to either HBFES LCE + Diet on an RT300 ergometer or Home-based (HB) Diet Alone intervention. Both groups will be routinely monitored via telemedicine while at home.

ELIGIBILITY:
Inclusion criteria:

* Adults 18-65 years of age (inclusive)
* Sex: male or female
* Women of child-bearing potential who agree to refrain from getting pregnant during the trial
* C4-T4 motor complete (AIS A&B) spinal cord injury for duration greater than 12 months
* <5% change in body weight over the past 12 months

Exclusion criteria:

* <22% body fat
* Unresponsive to neurostimulation
* Those who have participated in an FES or ACE exercise program (>60 minutes/week) within the past 3 months
* Known orthopaedic limitations
* Coronary artery disease
* Type 1 diabetes mellitus, insulin-requiring Type 2 or untreated diabetes mellitus (fasting glucose>126 or HgbA1c>7.0)
* Uncompensated Hypothyroidism (Stable on medication >1 year or not on medication)
* Renal disease
* Uncontrolled autonomic dysreflexia, recent (within 3 months)
* Deep vein thrombosis
* Pressure ulcers > Grade II
* Decisional impairment
* Any potential causes of autonomic dysreflexia at the discretion of the PI
* Prisoners
* Pregnant or nursing women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Tiozzo, PhD, MSCTI, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Home-Based Exercise & Diet Group | Home-Based Diet Alone Group
Started | 13 | 13
Completed | 10 | 12
Not Completed | 3 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Home-Based Exercise & Diet Group | Home-Based Diet Alone Group | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 11 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 14
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Injury duration [Mean (Standard Deviation); unit: years] | 5.5 (5.0) | 10.8 (8.4) | 8.2 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Percent Body Fat Assessed by DXA at Baseline and 21 Weeks
Description: Percent body fat will be assessed in percentage using Dual Energy x-ray absorbency (DXA). Assessments will be conducted at baseline and at 21 weeks to evaluate changes in body composition over time.
Time Frame: Baseline, 21 weeks
Population: Percent body fat was analyzed using DXA.
Measure: Mean (Standard Deviation); unit: % of body fat
Groups:
- Exercise and Diet: It included exercise (functional electrical stimulation leg cycling) and diet (nutrition counseling from a registered dietitian).
  The exercise group completed 3-5 remotely monitored weekly sessions, targeting ≥200 minutes of active exercise at 70% maximum heart rate. Dietary counseling was done weekly, one-on-one and it aimed to achieve a 200 kcal/day deficit from baseline energy intake.
- Diet Only: It included nutrition counseling from a registered dietitian (weekly and one-on-one), aiming to achieve a 200 kcal/day deficit from baseline energy intake.
Arm/Group | Exercise and Diet | Diet Only
Number analyzed (Participants) | 13 | 13
% of body fat
  Baseline | 26.6 (9.0) | 25.9 (9.6)
  21 weeks | 22.0 (5.3) | 25.6 (6.9)

2. Primary Outcome: Fat Free Mass
Description: Body composition will be assessed using Dual-Energy X-ray Absorptiometry (DXA), which provides precise measurements of both absolute fat mass (FM) and absolute fat-free mass (FFM) in kilograms. FFM represents a distinct component of total body mass and will be used to evaluate lean tissue (i.e.,FFM) over time.
Time Frame: Baseline, 21 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Home-Based Exercise & Diet Group | Home-Based Diet Alone Group
Number analyzed (Participants) | 13 | 13
kilograms
  Baseline | 48.7 (8.3) | 48.1 (6.8)
  21 weeks | 48.5 (7.1) | 49.4 (7.7)

3. Primary Outcome: Change in Insulin Sensitivity (Si)
Description: Insulin Sensitivity will be measured using intravenous glucose tolerance test (IVGTT)
Time Frame: Baseline, 21 weeks
Measure: Mean (Standard Deviation); unit: min^-1/microU/mL^-1) _x10^-4
Arm/Group | Home-Based Exercise & Diet Group | Home-Based Diet Alone Group
Number analyzed (Participants) | 13 | 13
min^-1/microU/mL^-1) _x10^-4
  Baseline | 4.1 (9.9) | 3.2 (4.3)
  21 weeks | 1.8 (1.5) | 1.5 (1.4)

4. Primary Outcome: Change in Glucose Effectiveness (Sg)
Description: Glucose Effectiveness will be measured using IVGTT
Time Frame: Baseline, 21 weeks
Measure: Mean (Standard Deviation); unit: glucose clearance per minute (min-¹)
Arm/Group | Home-Based Exercise & Diet Group | Home-Based Diet Alone Group
Number analyzed (Participants) | 13 | 13
glucose clearance per minute (min-¹)
  Baseline | 0.027 (0.016) | 0.019 (0.018)
  21 weeks | 0.027 (0.008) | 0.015 (0.006)

5. Primary Outcome: Change in Basal Metabolic Rate (BMR)
Description: BMR will be measured by indirect calorimetry
Time Frame: Baseline, 21 weeks
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Home-Based Exercise & Diet Group | Home-Based Diet Alone Group
Number analyzed (Participants) | 13 | 13
kcal/day
  Baseline | 1587.4 (249.5) | 1502.5 (234.6)
  21 weeks | 1588.8 (139.8) | 1510.0 (178.4)

6. Secondary Outcome: High Density Lipoprotein Cholesterol (HDL-C)
Description: HDL-C will be measured from blood serum samples
Time Frame: Baseline, 21 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Home-Based Exercise & Diet Group | Home-Based Diet Alone Group
Number analyzed (Participants) | 13 | 13
mg/dl
  Baseline | 40.4 (8.0) | 41.5 (12.4)
  21 weeks | 41.8 (7.4) | 39.7 (10.3)

7. Secondary Outcome: Change in Total Cholesterol : HDL-C Ratio
Description: Total Cholesterol HDL-C ratio will be calculated from blood serum samples reported as a numeric value, representing the ratio of Total Cholesterol to HDL-C.
Time Frame: Baseline, 21 weeks
Population: Ratio
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Exercise and Diet | Diet Only
Number analyzed (Participants) | 13 | 13
ratio
  Baseline | 4.66 (1.66) | 3.81 (1.30)
  21 weeks | 4.53 (1.46) | 3.95 (1.22)

8. Secondary Outcome: C-Reactive Protein (hsCRP)
Description: hsCRP will be measured from blood serum samples
Time Frame: Baseline, 21 weeks
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Exercise and Diet | Diet Only
Number analyzed (Participants) | 13 | 13
mg/L
  Baseline | 8.8 (12.4) | 8.8 (10.2)
  21 weeks | 2.6 (1.3) | 5.2 (4.0)

9. Secondary Outcome: Lower Extremity Bone Mineral Density (BMD) - Femur
Description: The changes in Bone Mineral Density will be measured using DXA scan
Time Frame: Baseline, 21 weeks
Measure: Mean (Standard Deviation); unit: g/cm³
Arm/Group | Home-Based Exercise & Diet Group | Home-Based Diet Alone Group
Number analyzed (Participants) | 13 | 13
g/cm³
  Baseline | 0.8 (0.1) | 0.7 (0.2)
  21 weeks | 0.8 (0.2) | 0.7 (0.2)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Home-Based Exercise & Diet Group | Home-Based Diet Alone Group
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 5/13 | 2/13
Other Adverse Events (participants affected / at risk) | 7/13 | 1/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home-Based Exercise & Diet Group (N=13) | Home-Based Diet Alone Group (N=13)
Heart failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (UTI) (Infections and infestations) | 1 (1) | 1 (1)
(Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Heterotopic ossification (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Cardiac disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Autonomic Dysreflexia (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home-Based Exercise & Diet Group (N=13) | Home-Based Diet Alone Group (N=13)
Skin Irritation (Skin and subcutaneous tissue disorders) | 7 (9) | 1 (1) — 7 participants had skin issues in exercise + diet group. However, 2 participants with skin issues in this group were unrelated to the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT03495986/Prot_SAP_001.pdf